CLINICAL TRIAL: NCT00402428
Title: Phase 3 Study to Evaluate the Efficacy and Safety of Albumin Interferon Alfa-2b in Combination With Ribavirin Compared With Peginterferon Alfa-2a in Combination With Ribavirin in Interferon Alfa Naive Subjects With CHC Genotype 1. ACHIEVE-1
Brief Title: Efficacy of Albumin Interferon Alfa-2b With Ribavirin Compared With Peg-IFN Alfa-2a With Ribavirin in IFN Naive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGS1008-C1060; ACHIEVE-1 (Other: Human Genome Sciences Inc.)
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Hepatitis C; CHC; HepC; Genotype 1; Hepatitis; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Hepatitis | interventions — peginterferon alfa-2a; Ribavirin

ARMS (3):
- 1 (Active Comparator): 180 mcg PEG-IFNx2a every 1 week (48 doses) + Ribavirin 1000 or 1200 mg/day
  Interventions: Drug: peginterferon alfa-2a; Drug: Ribavirin
- 2 (Experimental): 900 mcg alb-IFN every 2 weeks (24 doses)+ Ribavirin 1000 or 1200 mg/day
  Interventions: Drug: albumin interferon alfa-2b; Drug: Ribavirin
- 3 (Experimental): 1200 mcg alb-IFN every 2 weeks (24 doses)+ Ribavirin 1000 or 1200 mg/day
  Interventions: Drug: albumin interferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: albumin interferon alfa-2b — 900 mcg or 1200mcg every two week for 48 weeks
  Arms: 2; 3
Drug: peginterferon alfa-2a — 180 mcg once a week for 48 weeks
  Arms: 1
Drug: Ribavirin — 1000 mg/day(for subjects <75kg) or 1200 mg/day (for subjects
  =,> 75kg)

SUMMARY:
This is a phase 3, randomized, multi-center study to evaluate the efficacy and safety of albumin interferon alfa 2b (alb-IFN)in combination with ribavirin compared with peginterferon alfa-2a (PEGASYS or PEG-IFNa2a) in combination with ribavirin in subjects with chronic hepatitis C, genotype 1 who are IFNa treatment naive.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of chronic hepatitis C.
* Liver biopsy performed within 2 years of Day 0 or during screening.
* Infected with hepatitis C virus genotype 1.
* Interferon alfa treatment naïve (ie, have never been treated with an interferon product).
* Subjects are eligible to enter the study if they (or their partners) are not pregnant or nursing, are sterile, or of non childbearing potential, or are willing to practice abstinence or use appropriate birth control methods during the study and for 7 months after the last dose of ribavirin.
* Have compensated liver disease.

Key Exclusion Criteria:

* Decompensated liver disease including those subjects with a past history or presence of ascites, bleeding varices or hepatic encephalopathy.
* History of moderate, severe or uncontrolled psychiatric disease, especially depression, including a history of hospitalization or prior suicidal attempt.
* Positive for human immunodeficiency virus (HIV-1) or hepatitis B surface antigen (HBsAG).
* Clinical diagnosis of other causes of chronic liver disease including but not limited to hepatitis B, autoimmune hepatitis, primary biliary cirrhosis, alcoholic liver disease, hemochromatosis, Wilson's Disease, or alpha 1-antitrypsin deficiency.
* A history of immunologically mediated disease (eg, rheumatoid arthritis, inflammatory bowel disease, moderate/severe psoriasis, sarcoidosis, systemic lupus erythematosus).
* Active seizure disorder within the last 2 years.
* Organ transplant other than cornea and hair transplant.
* Clinically significant hemoglobinopathy (eg, thalassemia, sickle cell anemia).
* Cancer within the last 5 years(with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix).
* Drug or alcohol addiction within the last 6 months. Subjects in a supervised methadone treatment program may be enrolled in the study.
* Received any experimental agent within 28 days prior to Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1331 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | Week 72

SECONDARY OUTCOMES:
Rapid virologic response | Week 4
Early virologic response | Week 12
Undetectable HCV RNA | Week 24 and Week 48
Normalization of ALT (a liver enzyme) | Week 48
Quality of life evaluation | throughout the entire study
Safety assessments (physical exams, AE reporting, lab testing/analysis, HADS and Immunogenicity testing) | Throughout the entire study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (165):
- United States (65):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - UCSF Fresno, Fresno, California
  - Scripps Clinic, La Jolla, California
  - USC Keck School of Medicine, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA / West LA VAMC, Los Angeles, California
  - Huntington Medical Research Institutes, Pasadena, California
  - University California-San Diego, San Diego, California
  - San Diego Digestive Diseases Consultants, Inc, San Diego, California
  - VA San Diego Healthcare, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Colorado Health Sciences Ctr, Englewood, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Florida - Gainesville, Gainesville, Florida
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - Mayo Clinic Transplant Center, Jacksonville, Florida
  - Va Health Care System, Miami, Florida
  - University of Miami, Miami, Florida
  - Venture Research Institute, North Miami Beach, Florida
  - University Hepatitis Center, Sarasota, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - GI of Atlanta, Atlanta, Georgia
  - Northwest Georgia Gastroenterology Associates, Marietta, Georgia
  - Alan D Tice, MD, LLC, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiania University School of Medicine, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Center for Viral Hepatits, Baltimore, Maryland
  - Maryland Digestive Disease Center, Laurel, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Digestive Health Specialist, Tupelo, Mississippi
  - St. Louis University, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - New York Hospital - Cornell, New York, New York
  - Faculty Practice Associates, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Hospital of University of PA, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Nashville Gastroenterology, Nashville, Tennessee
  - Nashville Gastrointestinal Specialists, Nashville, Tennessee
  - Liver Institute at Methodist Dallas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwesten Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - GI & Liver Assoicates, Granbury, Texas
  - Liver Specialist of Texas, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - INOVA Fairfax Hospital, Annandale, Virginia
  - Metropolitan Research, Fairfax, Virginia
  - Virginia Commonwealth University Medical Ctr, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (16):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital Clinical School of Medicine University of New South Wales, Kogarah, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria, Victoria
  - Western Hospital, Footscray, Victoria
  - Austin Hospital, Heidelburg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth
- Austria (3):
  - Medizinische Universitätsklinik Graz, Graz
  - Univ.-Klinik fuer Innere Medizin, Innsbruck
  - Medical University of Vienna, Vienna
- Canada (11):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Manitoba Health Sciences Centre, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - University of Western Ontario Hospital, London, Ontario
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- Czechia (7):
  - Klinika infekcních chorob, Brno
  - Klinika Infekcních nemocí, Hradec Králové
  - Nemocnice s poliklinikou Melník, Mělník
  - Slezská nemocnice, Opava
  - Vseobecna fakultní nemocnice, Prague
  - Nuselská poliklinika, Prague
  - Ambulance pro interni a infekcni nemoci, Ústí nad Labem
- France (10):
  - Hopital Beaujon, Clichy
  - Hopital Henri Mondor, Créteil
  - CHU de Lyon, Hôpital de l'Hôtel Dieu, Lyon
  - Hopital Saint-Joseph, Marseille
  - Hopital de La Source, Orléans
  - Hôpital Saint-Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Haut-Leveque, Pessac
  - CHU Purpan Clinique Dieulafoy, Toulouse
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Germany (11):
  - UH Charite Berlin / Virchow Klinikum, Berlin
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Universitätsklinik Düsseldorf, Düsseldorf
  - UH Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main
  - Albert-Ludwigs-Universitaet Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Johannes Gutenberg-Universitaet Mainz, Mainz
  - Paracelsus Klinik der Stadt Marl, Marl
- India (3):
  - Dayanand Medical College and Hospital, Ludhiana
  - Jaslok Hospital and Research Centre and Breach Candy Hospital,, Mumbai
  - G.B.Pant Hospital, New Delhi
- Israel (6):
  - Bnei-Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Policlinico S.Orsola Malpighi, Bologna
  - IRCCS Ospedale Maggiore, Fondazione Policlinico Mangiagalli e Regina Elena, Università di Milano, Milan
  - Seconda Università di Napoli c/o Secondo Policlinico, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - I.R.C.C.S. Policlinico S. Matteo Università degli Studi di Pavia, Pavia
  - Casa Sollievo della Sofferenza IRCCS, San Giovanni Rotondo (FG)
  - Azienda Ospedaliera S. Giovanni Battista Molinette, Torino
- Poland (8):
  - Wojewódzki Szpital Specjalistyczny im.K. Dłuskiego, Bialystok
  - Szpital Specjalistyczny, Chorzów
  - Wojewódzki Szpital Zespolony, Kielce
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Uniwersytet Medyczny, Lodz
  - Akademia Medyczna, Warsaw
  - Wojewódzki Szpital Zaka?ny, Warsaw
  - Wojewódzki Szpital Specjalistyczny im. J. Gromkowskiego, Wroclaw
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico
- Romania (5):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Dr.Victor Babes, Bucharest
  - Spitalul Clinic de Adulti Cluj-Napoca, Cluj-Napoca
  - Institutul de Gastroenterologie si Hepatologie, Lasi
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona - Barcelona
  - Hopital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Carlos III, Madrid
  - Consorcio Hospital General Universitario de Valencia, Valencia
- United Kingdom (5):
  - Queen Elizabeth Medical Centre, Birmingham
  - Royal London Hospital, London
  - Imperial College London St Mary's Hospital Campus, London
  - Nottingham University Hospitals NHS Trust Queens Medical Centre Campus, Nottingham
  - Derriford Hospital, Plymouth

REFERENCES:
- [Background] Bain VG, Yoshida EM, Kaita KD, Swain MG, Heathcote EJ, Garcia A, Moore PA, Yu R, McHutchison JG, Subramanian GM. Dynamics of interferon-specific gene expression in peripheral blood of interferon alfa-naive patients with genotype 1 chronic hepatitis C infection treated with albumin-interferon alfa. Hepatol Res. 2006 Aug;35(4):256-62. doi: 10.1016/j.hepres.2006.04.005. Epub 2006 May 30. PMID 16731032
- [Background] Bain VG, Kaita KD, Yoshida EM, Swain MG, Heathcote EJ, Neumann AU, Fiscella M, Yu R, Osborn BL, Cronin PW, Freimuth WW, McHutchison JG, Subramanian GM. A phase 2 study to evaluate the antiviral activity, safety, and pharmacokinetics of recombinant human albumin-interferon alfa fusion protein in genotype 1 chronic hepatitis C patients. J Hepatol. 2006 Apr;44(4):671-8. doi: 10.1016/j.jhep.2005.12.011. Epub 2006 Jan 30. PMID 16487617
- [Background] S. Zeuzem, , Y. Benhamou, , D. Shouval, , V. Bain, S. Pianko, , R. Flisiak, , M. Grigorescu, , V. Rehak, , E. Yoshida, K. Kaita, , C. Hezode, A.U. Neumann, M. Subramanian, J. McHutchison. Interim (Week 12) Phase 2B Virological Efficacy and Safety Results of albumin interferon alfa-2b Combined with Ribavirin in Genotype 1 Chronic Hepatitis C Infection. EASL, 2006
- [Background] Vinod Rustgi, et al. A Dose-Escalation Study of albumin alfa-Ribavirin in Non-responders to Prior Interferon Based Therapy for Chronic Hepatitis C Infection Phase 2 Dose A Phase 2 Dose-Escalation Study of albumin interferon alfa interferon alfa-2b Combined with 2b Combined with Ribavirin in Non Non-responders to Prior Interferon. EASL, 2006
- [Background] Balan V, Nelson DR, Sulkowski MS, Everson GT, Lambiase LR, Wiesner RH, Dickson RC, Post AB, Redfield RR, Davis GL, Neumann AU, Osborn BL, Freimuth WW, Subramanian GM. A Phase I/II study evaluating escalating doses of recombinant human albumin-interferon-alpha fusion protein in chronic hepatitis C patients who have failed previous interferon-alpha-based therapy. Antivir Ther. 2006;11(1):35-45. PMID 16518958
- [Derived] Zeuzem S, Sulkowski MS, Lawitz EJ, Rustgi VK, Rodriguez-Torres M, Bacon BR, Grigorescu M, Tice AD, Lurie Y, Cianciara J, Muir AJ, Cronin PW, Pulkstenis E, Subramanian GM, McHutchison JG; ACHIEVE-1 Study Team. Albinterferon Alfa-2b was not inferior to pegylated interferon-alpha in a randomized trial of patients with chronic hepatitis C virus genotype 1. Gastroenterology. 2010 Oct;139(4):1257-66. doi: 10.1053/j.gastro.2010.06.066. Epub 2010 Jun 27. PMID 20600013